CLINICAL TRIAL: NCT05395546
Title: Digital Cognitive Behavioral Therapy (dCBT-I) for Maternal Insomnia During Pregnancy
Brief Title: Digital Cognitive Behavioral Therapy (dCBT-I) for Maternal Insomnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO2022-2213
Record Dates: First submitted 2022-05-16; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Digital Cognitive Behavioral Therapy for Insomnia (dCBT-I)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dCBT-I treatment group (Experimental)
  Interventions: Other: dCBT-I

INTERVENTIONS:
Other: dCBT-I — 1. Complete the evaluation of various scales and record a 7-day sleep diary before entering the group
  2. Receive a 6-week treatment after enrollment, insist on using the app every day (about 5-10 minutes), and receive regular follow-up from the project doctor
  3. Scale assessment needs to be completed at the end of treatment
  4. One month after the end of treatment, cooperate with relevant follow-up and complete the scale evaluation
  Other Names: Device: smartphone

SUMMARY:
Insomnia symptoms are common during pregnancy, especially in the second and third trimesters, which can reach more than 68%. Insomnia during pregnancy is not only associated with increased risk of preeclampsia, gestational diabetes, preterm labor, and cesarean section, but also increased postpartum poor sleep and postpartum depression. Cognitive behavioral therapy (CBT-I) and drug therapy for insomnia are the two main methods of insomnia treatment. Drug therapy is the more commonly used traditional treatment method, but there may be certain drug risks. Therefore, non-drug methods for Insomnia in pregnant women is much safer.

Cognitive-behavioral therapy for insomnia is a psychological therapy for insomnia. Compared with sedative-hypnotic drugs, its therapeutic effect is slow, but the curative effect is long-lasting, with less relapse after treatment and no invasive side effects. Multiple guidelines recommend it as first-line therapy for insomnia. And "Digital Cognitive Behavioral Therapy" (dCBT-I), is based on CBT-I, a therapy provided by the Internet and smartphones, which simulates face-to-face CBT-I in reality. It can provide more convenient medical services for the special group of pregnant women, improve sleep, improve mental symptoms, life treatment, and reduce the risk of adverse outcomes for mothers and children.

The Womens' Hospital, Zhejiang University School of Medicine is conducting a clinical study on "Digital Cognitive Behavioral Therapy (dCBT-I) for maternal Insomnia during pregnancy". The primary goal of this research project was to examine the efficacy of dCBT-I ("RuMian") in the treatment of maternal insomnia. "RuMian" is a fully automatic dCBT-I application developed in China, and subjects will use it for free.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years old
* 20-32 weeks of pregnancy, singleton pregnancy and regular obstetric examination at Zhejiang University Women's Hospital
* There has been a high frequency of insomnia symptoms
* According to the preliminary assessment by the project team, it meets the diagnostic criteria for insomnia
* Possess a smart phone and can operate it proficiently, with normal reading and writing comprehension ability, clear consciousness, and able to cooperate with the research to complete the questionnaire independently.

Exclusion Criteria:

* Assess the risk of preterm birth and concurrent pregnancy-related diseases;
* Completion of the 7-day sleep diary in the baseline period < 4 days;
* Combined with severe anxiety/depression;
* Suicidal tendencies or severe mental illness (bipolar disorder, schizophrenia, paranoid psychosis, etc.);
* Edinburgh Pregnancy Depression Scale (EPDS) total score ≥ 15;
* Have drug dependence or have taken anti-anxiety, anti-depression, sedative or hypnotic drugs for mental diseases within the past 3 months;
* Participated in interventions such as meditation courses, childbirth yoga or cognitive behavioral therapy in the past 1 year;
* Complicated with serious physical diseases such as heart failure and tumor;
* Combined with sleep disorders such as severe obstructive sleep apnea that require further evaluation and treatment;
* There is alcohol and cigarette dependence;
* Shift work;
* Severe visual or hearing impairment and unable to use mobile phones normally;
* Physical illness with unstable condition, or illness itself that may interfere with cognitive behavioral therapy for insomnia.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-07-15 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Change of "Insomnia Severity Index(ISI)" | From before treatment to the end of treatment (an average of 42 days)
  Insomnia Severity Index(ISI),the minimum and maximum values are 0 and 28, and higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change of "Pittsburgh Sleep Quality Index（PSQI）" | From before treatment to the end of treatment (an average of 42 days)
  Pittsburgh Sleep Quality Index（PSQI）,the minimum and maximum values are 0 and 21, and higher scores mean a worse outcome.
Change of "sleep onset latency（SOL）" | From before treatment to the end of treatment (an average of 42 days)
  simple questionnaire will be used to assess this outcome of sleep onset latency（SOL）
Change of "wake up after sleep onset(WASO)" | From before treatment to the end of treatment (an average of 42 days)
  simple questionnaire will be used to assess this outcome of WASO
Change of "sleep efficiency（SE）" | From before treatment to the end of treatment (an average of 42 days)
  combination of questionnaire and calculate will be used to assess this outcome of SE
Change of "Number of wake ups during the night" | From before treatment to the end of treatment (an average of 42 days)
  Number of wake ups during the night
Change of "total sleep time（TST）" | From before treatment to the end of treatment (an average of 42 days)
  total sleep time（TST）
Change of "Edinburgh Pregnancy Depression Scale（EPDS）" | From before treatment to the end of treatment (an average of 42 days)
  Edinburgh Pregnancy Depression Scale（EPDS）,the minimum and maximum values are 0 and 30, and higher scores mean a worse outcome.
Change of "Self-rating Anxiety Scale（SAS）" | From before treatment to the end of treatment (an average of 42 days)
  Self-rating Anxiety Scale（SAS）, the minimum and maximum values are 25 and 100, and higher scores mean a worse outcome.